CLINICAL TRIAL: NCT04165057
Title: Efficacy and Safety of Optimal Muscle Tension Management During Laparoscopic Cholecystectomy - a Prospective Randomized Control Study
Brief Title: Efficacy and Safety of Optimal Muscle Tension Management During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108-084-F
Record Dates: First submitted 2019-11-03; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia
Keywords: Laparoscopic surgery; Optimal muscle tension; Neuromuscular monitoring; Neuromuscular blockade; Sugammadex

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group OMT (Active Comparator): Optimal muscle tension management
  Interventions: Other: Optimal muscle tension management
- Group Control (No Intervention): Conventional anesthetic management

INTERVENTIONS:
Other: Optimal muscle tension management — including TOF monitor and reversal of neuromuscular blockade agent : sugammadex
  Arms: Group OMT

SUMMARY:
Our study is intended to compare optimal muscle tension management or conventional anesthetic management in laparoscopic cholecystectomy about surgical condition during the surgery and other conditions after surgery at POR.

DETAILED DESCRIPTION:
This study is intended to recruit 70 patients undergoing laparoscopic cholecystectomy, whom will be randomized to receive optimal muscle tension management or conventional anesthetic management without optimal muscle tension management. Our primary hypothesis is that optimal muscle tension management provides improved surgical conditions and less intra-abdominal pressure required. The secondary endpoints include surgical duration, intraoperative complications, total amount of muscle relaxants, respiratory and hemodynamic changes during surgery, extubation time and any events during post-anesthetic recovery.

ELIGIBILITY:
Inclusion Criteria:

* age 20~80 years old
* ASA score : 1-2
* Regular laparoscopic cholecystectomy

Exclusion Criteria:

* Renal function impairement (eGFR < 60 ml/min/1.73m2) or ESRD
* BMI < 18.5 kg/m2 or >30 kg/m2
* History of other abdominal surgery
* Allergy to rocuronium, cisatracurium, neostigmine or sugammadex
* Emergent surgery
* Convert to open cholecystectomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical condition | 5 minutes
  Surgeon describe CO2 inflation condition by 4 point King Score (1-4).
  1. excellent
  2. good
  3. acceptable
  4. poor or unacceptable

SECONDARY OUTCOMES:
Peak inspiratory pressure during surgery | 1 hour
  Peak inspiratory pressure during surgery
Mean blood pressure | Every 5 mins
  Mean blood pressure during the CO2 inflation
Total surgical time | 1 hour
  Total surgical time
Total Rocuronium doses during surgery | 1 hour
  Total Rocuronium doses during surgery
Pain score at Postoperative room | 1 hour
  describe by 11 points Numeric rating scales (0-10). From 0 which means "no pain" to 10 means "worst pain"
Heart Rate | every 5 mins
  Every beat per minutes heart rate during CO2 inflation
Respiratory complications | Every 5 mins
  Record any respiratory complications including desaturations (<95%, more than 30 seconds, Rispiratory rate < 8), aspiration or airway obstruction

CONTACTS AND LOCATIONS:
Overall Officials: MING-HUI HUNG, MD, Study Director — National Taiwan University Hospital Hsinchu Branch
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No